CLINICAL TRIAL: NCT00790023
Title: A Randomized, Multicenter, Double Blind, Placebo Controlled, Parallel Group, Phase III Clinical Trial to Assess the Efficacy and Safety of Ciclesonide HFA Nasal Aerosol (160 μg Once Daily and 80 μg Once Daily) for the Treatment of Seasonal Allergic Rhinitis (SAR) to Mountain Cedar in Subjects 12 Years and Older.
Brief Title: Clinical Trial to Assess the Efficacy and Safety of Ciclesonide Hydrofluoroalkane (HFA) Nasal Aerosol for the Treatment of Seasonal Allergic Rhinitis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sumitomo Pharma America, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 060-622
Record Dates: First submitted 2008-11-11; First posted 2008-11-13 (Estimated); Results first posted 2012-06-08 (Estimated); Last update posted 2016-04-08 (Estimated); Status verified 2016-03

CONDITIONS: Seasonal Allergic Rhinitis
Keywords: SAR
MeSH Terms: conditions — Rhinitis, Allergic, Seasonal | interventions — ciclesonide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- 80 mcg Ciclesonide (Experimental): 80 mcg Ciclesonide once daily
  Interventions: Drug: 80 mcg Ciclesonide
- 160 mcg Ciclesonide (Experimental): 160 mcg Ciclesonide once daily
  Interventions: Drug: 160 mcg Ciclesonide
- Placebo (Placebo Comparator): Placebo once daily
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: 80 mcg Ciclesonide — 80 mcg Ciclesonide HFA Inhaler once daily (one actuation per nostril)
  Arms: 80 mcg Ciclesonide
Drug: 160 mcg Ciclesonide — 160 mcg Ciclesonide HFA Inhaler once daily (one actuation per nostril)
  Arms: 160 mcg Ciclesonide
Drug: Placebo — Placebo HFA Inhaler once daily (one actuation per nostril)
  Arms: Placebo

SUMMARY:
To demonstrate the efficacy of ciclesonide HFA applied as a nasal aerosol (160 μg and 80 μg) once daily compared to placebo in subjects with SAR.

DETAILED DESCRIPTION:
This is a randomized, double blind, placebo controlled, parallel group, multicenter study to demonstrate the efficacy of ciclesonide HFA applied as a nasal aerosol (160 μg and 80 μg) once daily compared to placebo in subjects with SAR. This study was previously posted by Sepracor Inc. In October 2009, Sepracor Inc. was acquired by Dainippon Sumitomo Pharma., and in October 2010, Sepracor Inc's name was changed to Sunovion Pharmaceuticals Inc.

ELIGIBILITY:
Inclusion Criteria:

* Give written informed consent, including privacy authorization as well as adherence to concomitant medication withholding periods, prior to participation.
* Male or female 12 years and older, as of the Screening Visit (Visit 1).
* Subject must be in general good health (defined as the absence of any clinically relevant abnormalities as determined by the Investigator) based on screening physical examination, medical history, and clinical laboratory values (Hematology, Chemistries and Urinalysis).
* A history of SAR to Mountain Cedar for a minimum of two years immediately preceding the study Screening Visit (Visit 1). The SAR must have been of sufficient severity to have required treatment (either continuous or intermittent) in the past and in the Investigator's judgment (through exposure to allergen) is expected to require treatment throughout the entire study period.
* A demonstrated sensitivity to Mountain Cedar known to induce SAR through a standard skin prick test administered at Visit 1 (screening). A positive test is defined as a wheal diameter at least 5 mm larger than the control wheal (normal saline) for the skin prick test.
* Subject, if female 65 years of age or younger, must have a negative serum pregnancy test (performed at Visit 1) prior to randomization at Visit 2. Women of childbearing potential (excluding females at least two years postmenopausal or surgically sterile) must sign the Women of Childbearing Potential Addendum to the informed consent form. Females of childbearing potential must be instructed to and agree to avoid pregnancy during the study and must use an acceptable method of birth control:

  1. An oral contraceptive, an intrauterine device (IUD), implantable contraceptive, transdermal or injectable contraceptive for at least 1 month prior to entering the study and will continue its use throughout the study and for thirty days following study participation.
  2. Barrier method of contraception, eg, condom and/or diaphragm with spermicide while participating in the study.
  3. Abstinence.
* Subject or parent/guardian must possess an educational level and degree of understanding of English that enables them to communicate suitably with the Investigator and study coordinator as well as accurately complete both the AR diary and RQLQ(S).

Exclusion Criteria:

* Female subject who is pregnant or lactating.
* History of physical findings of nasal pathology, including nasal polyps or other clinically significant respiratory tract malformations; recent nasal biopsy; nasal trauma; nasal ulcers or perforations; or surgery and atrophic rhinitis or rhinitis medicamentosa (all within the last 60 days prior to the Screening Visit).
* Participation in any investigational drug trial within the 30 days preceding the Screening Visit (Visit 1) or planned participation in another investigational drug trial at any time during this trial.
* A known hypersensitivity to any corticosteroid or any of the excipients in the formulation of ciclesonide.
* History of a respiratory infection or disorder [including, but not limited to bronchitis, pneumonia, chronic sinusitis, influenza, severe acute respiratory syndrome (SARS)] within the 14 days preceding the Screening Visit (Visit 1).
* History of alcohol or drug abuse (or a positive urine drug screen at Visit 1) within two years preceding the Screening Visit.
* History of a positive test for HIV, hepatitis B or hepatitis C.
* Plans to travel outside the study area (the known pollen area for the investigative site) for more than 24 hours during the Run in period.
* Plans to travel outside the study area (the known pollen area for the investigative site) for 2 or more consecutive days between Randomization Visit (Visit 3) and the final Treatment Visit (Visit 5).
* Active asthma requiring treatment with inhaled or systemic corticosteroids and/or routine use of beta agonists and any controller drugs (e.g., theophylline, leukotriene antagonists, etc.); intermittent use (less than or equal to 3 uses per week) of inhaled short acting beta-agonists is acceptable.
* Use of any prohibited concomitant medications within the prescribed (per protocol) time period prior to the Screening Visit and expected use during treatment period.
* Use of antibiotic therapy for acute conditions within 14 days prior to the Screening Visit. Low doses of antibiotics taken for prophylaxis are permitted if the therapy was started prior to the Screening Visit and is expected to continue throughout the trial.
* Initiation of immunotherapy during the study period or dose escalation during the study period. However, initiation of immunotherapy 90 days or more prior to the Screening Visit and use of a stable (maintenance) dose (30 days or more) may be considered for inclusion.
* Previous participation in an intranasal ciclesonide HFA nasal aerosol study.
* Non-vaccinated exposure to or active infection with, chickenpox or measles within the 21 days preceding the Screening Visit.
* Use of topical corticosteroids in concentrations in excess of 1% hydrocortisone or equivalent within 30 days prior to Visit 2; use of a topical hydrocortisone or equivalent in any concentration covering greater than 20% of the body surface; or presence of an underlying condition (as judged by the investigator) that can reasonably be expected to require treatment with such preparations during the course of the study.
* Initiation of pimecrolimus cream 1% or greater or tacrolimus ointment 0.03% or greater during the study period or planned dose escalation during the study period. However, initiation of these creams/ointments 30 days or more prior to the Visit 1 and use of a stable (maintenance) dose during the study period may be considered for inclusion.
* Study participation by clinical investigator site employees and/or their immediate relatives.
* Study participation by more than one subject from the same household at the same time.
* Have any of the following conditions that are judged by the investigator to be clinically significant and/or affect the subject's ability to participate in the clinical trial: impaired hepatic function including alcohol-related liver disease or cirrhosis;

  * history of ocular disturbances e.g. glaucoma or posterior subcapsular cataracts;
  * any systemic infection;
  * hematological, hepatic, renal, endocrine (except for controlled diabetes mellitus or postmenopausal symptoms or hypothyroidism);
  * gastrointestinal disease;
  * malignancy (excluding basal cell carcinoma);
  * current neuropsychological condition with or without drug therapy.
* Any condition that, in the judgment of the investigator, would preclude the subject from completing the protocol with capture of the assessments as written.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 707 (Actual)
Dates: Start 2008-11; Primary Completion 2009-02 (Actual); Study Completion 2009-02 (Actual)

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - Austin, Texas
  - Kerrville, Texas
  - New Braunfels, Texas
  - San Antonio, Texas

REFERENCES:
- [Result] Ratner P, Jacobs R, Mohar D, Huang H, Desai SY, Hinkle J. Evaluation of the efficacy and safety of ciclesonide hydrofluoroalkane nasal aerosol, 80 or 160 mug once daily, for the treatment of seasonal allergic rhinitis. Ann Allergy Asthma Immunol. 2010 Dec;105(6):471-9. doi: 10.1016/j.anai.2010.09.024. PMID 21130386

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | 80 mcg Ciclesonide | 160 mcg Ciclesonide | Placebo
Started | 237 | 235 | 235
Completed | 226 | 225 | 214
Not Completed | 11 | 10 | 21
Not completed — Adverse Event | 2 | 1 | 4
Not completed — Protocol Violation | 2 | 4 | 2
Not completed — Withdrawal by Subject | 2 | 0 | 6
Not completed — Lost to Follow-up | 0 | 0 | 1
Not completed — Other | 5 | 5 | 8

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 80 mcg Ciclesonide | 160 mcg Ciclesonide | Placebo | Total
Number analyzed (Participants) | 237 | 235 | 235 | 707
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 11 | 8 | 12 | 31
  Between 18 and 65 years | 220 | 217 | 203 | 640
  >=65 years | 6 | 10 | 20 | 36
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.1 (12.7) | 42.1 (12.9) | 42.2 (13.9) | 41.8 (13.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 159 | 155 | 155 | 469
  Male | 78 | 80 | 80 | 238
Race/Ethnicity, Customized [Number; unit: participants]
  White/Caucasian | 218 | 220 | 220 | 658
  Black/African American | 13 | 8 | 14 | 35
  Asian | 4 | 3 | 1 | 8
  American Indian or Alaska Native | 0 | 2 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 2 | 0 | 2
  Multiple | 2 | 0 | 0 | 2
Baseline reflective total nasal symptom score (rTNSS) [Mean (Standard Deviation); unit: Units on a scale] — TNSS is the sum of individual symptoms of runny nose, sneezing, itchy nose, and nasal congestions. Subjects assess each individual symptoms on a scale of 0-3 where:
  0 = absent
  1. = mild
  2. = moderate
  3. = severe. Therefore, rTNSS values range from 0-12 (with 0 representing an absence of symptoms and higher scores reflecting more severe symptoms). Reflective TNSS measures these symptoms over the previous 12-hour time interval. Baseline was the average of the AM and PM responses obtained during the run-in period up to 6 days prior to randomization.
  Units on a scale
    AM | 9.36 (1.76) | 9.47 (1.68) | 9.08 (1.85) | 9.31 (1.77)
    PM | 9.28 (1.92) | 9.44 (1.80) | 9.13 (1.87) | 9.28 (1.87)
    AM and PM | 9.32 (1.77) | 9.46 (1.67) | 9.10 (1.80) | 9.29 (1.75)
Baseline instantaneous total nasal symptom score (iTNSS) [Mean (Standard Deviation); unit: Units on a scale] — TNSS is the sum of individual symptoms of runny nose, sneezing, itchy nose, and nasal congestions. Subjects assess each individual symptoms on a scale of 0-3 where:
  0 = absent
  1. = mild
  2. = moderate
  3. = severe. Therefore, iTNSS values range from 0-12 (with 0 representing an absence of symptoms and higher scores reflecting more severe symptoms). Instantaneous TNSS measures these symptoms over the previous 10 minute time interval. Baseline was the average of the AM and PM responses obtained during the run-in period up to 6 days prior to randomization.
  Units on a scale
    AM | 8.83 (2.03) | 9.05 (2.02) | 8.74 (2.05) | 8.87 (2.03)
    PM | 8.53 (2.22) | 8.82 (2.14) | 8.48 (2.21) | 8.61 (2.19)
    AM and PM | 8.68 (2.05) | 8.94 (2.00) | 8.61 (2.06) | 8.74 (2.04)
Baseline reflective total ocular symptom score (rTOSS) in subjects with (rTOSS) ≥5.0 [Mean (Standard Deviation); unit: Units on a scale] — Total Ocular Symptom Score(TOSS) is the sum of individual ocular symptoms of itching, tearing, and redness. Subjects assess each individual symptoms on a scale of 0-3 where:
  0 = absent
  1. = mild
  2. = moderate
  3. = severe Therefore, TOSS ranges from 0-9 (with 0 representing an absence of symptoms and higher scores reflecting more severe symptoms). Reflective TOSS symptom scores assess symptoms over the previous 12-hour time interval. Baseline was the average of the AM and PM responses obtained during the run-in period up to 6 days prior to randomization.
  Units on a scale
    AM | 6.89 (1.27) | 6.98 (1.22) | 6.95 (1.33) | 6.94 (1.27)
    PM | 6.90 (1.24) | 7.04 (1.13) | 6.96 (1.25) | 6.97 (1.21)
    AM and PM | 6.89 (1.19) | 7.01 (1.11) | 6.95 (1.23) | 6.95 (1.18)
Baseline instantaneous total ocular symptom score (iTOSS) in subjects with (iTOSS) ≥5.0 [Mean (Standard Deviation); unit: Units on a scale] — TOSS is the sum of individual ocular symptoms of itching, tearing, and redness. Subjects assess each individual symptoms on a scale of 0-3 where:
  0 = absent
  1. = mild
  2. = moderate
  3. = severe Therefore, TOSS ranges from 0-9 (with 0 representing an absence of symptoms and higher scores reflecting more severe symptoms). Instantaneous TOSS symptom scores assess symptoms over the previous 10 minute time interval. Baseline was the average of the AM and PM responses obtained during the run-in period up to 6 days prior to randomization.
  Units on a scale
    AM | 6.91 (1.19) | 7.04 (1.16) | 7.17 (1.19) | 7.03 (1.18)
    PM | 6.67 (1.29) | 6.81 (1.24) | 6.86 (1.35) | 6.78 (1.29)
    AM and PM | 6.79 (1.14) | 6.92 (1.11) | 7.01 (1.19) | 6.90 (1.15)
Baseline reflective nasal symptom score (rNSS) [Mean (Standard Deviation); unit: Units on a scale] — NSS is the assessment of the individual symptoms of runny nose, sneezing, itchy nose, and nasal congestions. Subjects assess each individual symptoms on a scale of 0-3 where:
  0 = absent
  1. = mild
  2. = moderate
  3. = severe Reflective NSS measures these symptoms over the previous 12-hour time interval. Baseline was the average of the AM and PM responses obtained during the run-in period up to 6 days prior to randomization.
  Units on a scale
    AM Sneezing | 2.02 (0.73) | 2.11 (0.62) | 2.00 (0.71) | 2.04 (0.69)
    AM Runny Nose | 2.44 (0.55) | 2.41 (0.56) | 2.37 (0.57) | 2.41 (0.56)
    AM Nasal Itching | 2.33 (0.59) | 2.35 (0.54) | 2.22 (0.61) | 2.30 (0.58)
    AM Nasal Congestion | 2.57 (0.43) | 2.60 (0.43) | 2.48 (0.50) | 2.55 (0.46)
    PM Sneezing | 2.08 (0.69) | 2.17 (0.61) | 2.11 (0.64) | 2.12 (0.65)
    PM Runny Nose | 2.39 (0.59) | 2.39 (0.58) | 2.35 (0.58) | 2.38 (0.58)
    PM Nasal Itching | 2.32 (0.61) | 2.36 (0.54) | 2.25 (0.62) | 2.31 (0.59)
    PM Nasal Congestion | 2.49 (0.51) | 2.52 (0.48) | 2.42 (0.53) | 2.48 (0.51)
    AM and PM Sneezing | 2.05 (0.69) | 2.14 (0.59) | 2.05 (0.65) | 2.08 (0.65)
    AM and PM Runny Nose | 2.41 (0.55) | 2.40 (0.55) | 2.36 (0.56) | 2.39 (0.55)
    AM and PM Nasal Itching | 2.32 (0.58) | 2.36 (0.53) | 2.23 (0.59) | 2.30 (0.57)
    AM and PM Nasal Congestion | 2.53 (0.44) | 2.56 (0.43) | 2.45 (0.50) | 2.51 (0.46)
Baseline instantaneous nasal symptom score (iNSS) [Mean (Standard Deviation); unit: Units on a scale] — NSS is the assessment of the individual symptoms of runny nose, sneezing, itchy nose, and nasal congestions. Subjects assess each individual symptoms on a scale of 0-3 where: 0 = absent (no sign/symptom evident);
  1. = mild
  2. = moderate
  3. = severe Instantaneous NSS measures these symptoms over the previous 10 minute time interval. Baseline was the average of the AM and PM responses obtained during the run-in period up to 6 days prior to randomization.
  Units on a scale
    AM Sneezing | 1.72 (0.91) | 1.83 (0.83) | 1.77 (0.89) | 1.77 (0.88)
    AM Runny Nose | 2.35 (0.59) | 2.35 (0.64) | 2.32 (0.61) | 2.34 (0.61)
    AM Nasal Itching | 2.26 (0.62) | 2.30 (0.61) | 2.18 (0.61) | 2.24 (0.62)
    AM Nasal Congestion | 2.50 (0.48) | 2.58 (0.48) | 2.47 (0.52) | 2.52 (0.49)
    PM Sneezing | 1.77 (0.85) | 1.92 (0.79) | 1.81 (0.86) | 1.83 (0.84)
    PM Runny Nose | 2.23 (0.66) | 2.26 (0.66) | 2.23 (0.63) | 2.24 (0.65)
    PM Nasal Itching | 2.17 (0.67) | 2.24 (0.64) | 2.11 (0.66) | 2.17 (0.66)
    PM Nasal Congestion | 2.36 (0.57) | 2.39 (0.53) | 2.33 (0.57) | 2.36 (0.55)
    AM and PM Sneezing | 1.75 (0.86) | 1.88 (0.78) | 1.79 (0.85) | 1.80 (0.83)
    AM and PM Runny Nose | 2.29 (0.60) | 2.30 (0.62) | 2.27 (0.59) | 2.29 (0.60)
    AM and PM Nasal Itching | 2.21 (0.62) | 2.27 (0.60) | 2.15 (0.61) | 2.21 (0.61)
    AM and PM Nasal Congestion | 2.43 (0.49) | 2.49 (0.47) | 2.40 (0.52) | 2.44 (0.49)
Baseline individual reflective ocular symptom score (rOSS) in subjects with (rTOSS) ≥5.0 [Median (Standard Deviation); unit: Units on a scale] — OSS is the assessment of the individual symptoms of runny nose, sneezing, itchy nose, and nasal congestions. Subjects assess each individual symptoms on a scale of 0-3 where:
  0 = absent
  1. = mild
  2. = moderate
  3. = severe Reflective OSS measures these symptoms over the previous 12-hour time interval. Baseline was the average of the AM and PM responses obtained during the run-in period up to 6 days prior to randomization. rTOSS values range from 0-12 (with 0 representing an absence of symptoms and higher scores reflecting more severe symptoms).
  Units on a scale
    AM Itching Eyes | 2.48 (0.42) | 2.45 (0.50) | 2.42 (0.49) | 2.45 (0.47)
    AM Redness of Eyes | 2.14 (0.59) | 2.26 (0.53) | 2.25 (0.55) | 2.22 (0.56)
    AM Tearing Eyes | 2.26 (0.52) | 2.27 (0.48) | 2.27 (0.53) | 2.27 (0.51)
    PM Itching of Eyes | 2.47 (0.40) | 2.48 (0.43) | 2.42 (0.45) | 2.46 (0.43)
    PM Redness of Eyes | 2.15 (0.57) | 2.25 (0.50) | 2.28 (0.55) | 2.22 (0.54)
    PM Tearing Eyes | 2.28 (0.50) | 2.31 (0.46) | 2.26 (0.50) | 2.28 (0.48)
    AM and PM Itching Eyes | 2.48 (0.39) | 2.47 (0.44) | 2.42 (0.45) | 2.46 (0.42)
    AM and PM Redness of Eyes | 2.14 (0.56) | 2.25 (0.50) | 2.27 (0.53) | 2.22 (0.53)
    AM and PM Tearing Eyes | 2.27 (0.48) | 2.29 (0.44) | 2.26 (0.49) | 2.27 (0.47)
Baseline individual instantaneous ocular symtom score (iOSS) in subjects with (iTOSS) ≥5.0 [Mean (Standard Deviation); unit: Units on scale] — OSS is the assessment of the individual symptoms of runny nose, sneezing, itchy nose, and nasal congestions. Subjects assess each individual symptoms on a scale of 0-3 where:
  0 = absent
  1. = mild
  2. = moderate
  3. = severe Instantaneous OSS measures these symptoms over the previous 10 minute time interval. Baseline was the average of the AM and PM responses obtained during the run-in period up to 6 days prior to randomization. rTOSS values range from 0-12 (with 0 representing an absence of symptoms and higher scores reflecting more severe symptoms).
  Units on scale
    AM Itching Eyes | 2.44 (0.44) | 2.44 (0.46) | 2.48 (0.45) | 2.45 (0.45)
    AM Redness of Eyes | 2.22 (0.56) | 2.32 (0.51) | 2.36 (0.52) | 2.30 (0.53)
    AM Tearing Eyes | 2.25 (0.50) | 2.27 (0.48) | 2.33 (0.54) | 2.28 (0.51)
    PM Itching Eyes | 2.38 (0.41) | 2.40 (0.47) | 2.39 (0.49) | 2.39 (0.46)
    PM Redness of Eyes | 2.12 (0.58) | 2.22 (0.52) | 2.28 (0.55) | 2.20 (0.55)
    PM Tearing Eyes | 2.17 (0.52) | 2.19 (0.49) | 2.19 (0.56) | 2.18 (0.52)
    AM and PM Itching Eyes | 2.41 (0.38) | 2.42 (0.43) | 2.43 (0.45) | 2.42 (0.42)
    AM and PM Redness of Eyes | 2.17 (0.54) | 2.27 (0.49) | 2.32 (0.51) | 2.25 (0.51)
    AM and PM Tearing Eyes | 2.21 (0.47) | 2.23 (0.45) | 2.26 (0.51) | 2.23 (0.47)
Baseline Instantaneous Total Ocular Symptoms Scores (iTOSS)] for Onset of Nasal Improvement [Mean (Standard Deviation); unit: Hours] — Baseline is the last non-missing instantaneous AM assessment on or before Day 1. Onset of nasal improvement is defined as the first assessment at which instantaneous TNSS for active treatment demonstrates an improvement over placebo from baseline with one-sided p-value of <= 0.025.
  Hours | 6.85 (1.72) | 7.02 (1.54) | 6.98 (1.60) | 6.95 (1.62)
Baseline Rhinoconjunctivitis Quality of Life Questionnaire (RQLQ) in subject with RQLQ(S) score ≥3. [Mean (Standard Deviation); unit: units on a scale] — RQLQ(S)consists of 28 questions, each question measured on a scale of 0-6 where a higher score indicates poor quality of life. Domains: Activities (questions 1-3), Sleep (questions 4-6), Non-Nose/Eye Symptoms (questions 7-13), Practical Problems (questions 14-16), Nasal Symptoms (questions 17-20), Eye Symptoms (questions 21-24), and Emotional (questions 25-28). The overall RQLQ(S) score was calculated as the average of the mean domain scores.
  units on a scale | 4.52 (0.77) | 4.49 (0.78) | 4.43 (0.83) | 4.48 (0.79)
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 109 | 102 | 109 | 320
  Not Hispanic or Latino | 128 | 133 | 126 | 387

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Daily Subject-reported AM and PM Reflective Total Nasal Symptom Score (rTNSS) Averaged Over the Two-week Treatment Period.
Description: TNSS is the sum of individual symptoms of runny nose, sneezing, itchy nose, and nasal congestions. Subjects assess each individual symptoms on a scale of 0-3 where:
  0 = absent
  1. = mild
  2. = moderate
  3. = severe Therefore, rTNSS values range from 0-12 (with 0 representing an absence of symptoms and higher scores reflecting more severe symptoms). Reflective TNSS measures these symptoms over the previous 12-hour time interval. Difference was calculated as the two week treatment average - baseline. Greater reductions in the change from baseline score indicate greater improvement.
Time Frame: Week 0-2
Population: Intent to treat population.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | 80 mcg Ciclesonide | 160 mcg Ciclesonide | Placebo
Number analyzed (Participants) | 237 | 234 | 234
units on a scale | -1.45 (0.14) | -1.59 (0.14) | -0.51 (0.14)
Statistical Analysis 1: Comparison: 80 mcg Ciclesonide vs Placebo; The null hypothesis is that there is no difference in primary outcome when compare active to placebo group. The alternative hypothesis is that there is a difference in primary outcome when compare active to placebo group. It was estimated that 200 subjects per group will provide at least 85% power to detect a difference between treatment groups of 0.7 in the change from baseline in rTNSS with a two-sided alpha level of 0.025; Test type: Superiority or Other; p < 0.0001, ANCOVA — The p-value from primary outcome was adjusted at alpha=0.025; Mean Difference (Final Values) = 0.94, 95% CI 2-sided [0.57 to 1.32]
Statistical Analysis 2: Comparison: 160 mcg Ciclesonide vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.0001, ANCOVA — The p-value from primary outcome was adjusted at alpha=0.025; Mean Difference (Final Values) = 1.08, 95% CI 2-sided [0.70 to 1.45]

2. Secondary Outcome: Change From Baseline in Daily Subject-reported AM and PM iTNSS Averaged Over the Two-week Treatment Period.
Description: TNSS is the sum of individual symptoms of runny nose, sneezing, itchy nose, and nasal congestions. Subjects assess each individual symptoms on a scale of 0-3 where:
  0 = absent
  1. = mild
  2. = moderate
  3. = severe Therefore, rTNSS values range from 0-12 (with 0 representing an absence of symptoms and higher scores reflecting more severe symptoms). Instantaneous TNSS measures these symptoms over the previous 10 minute time interval. Difference was calculated as the two week treatment average - baseline. Greater reductions in the change from baseline score indicate greater improvement.
Time Frame: Week 0-2
Population: Intent to treat population
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | 80 mcg Ciclesonide | 160 mcg Ciclesonide | Placebo
Number analyzed (Participants) | 237 | 234 | 234
units on a scale | -1.34 (0.13) | -1.47 (0.13) | -0.47 (0.13)
Statistical Analysis 1: Comparison: 80 mcg Ciclesonide vs Placebo; Dmitrienko's tree-structured gatekeeping method was used for multiple comparisons; Test type: Superiority or Other; p < 0.0001, ANCOVA; Mean Difference (Final Values) = 0.87, 95% CI 2-sided [0.50 to 1.25]
Statistical Analysis 2: Comparison: 160 mcg Ciclesonide vs Placebo; Dmitrienko's tree-structured gatekeeping method was used for multiple comparisons; Test type: Superiority or Other; p < 0.0001, ANCOVA; Mean Difference (Final Values) = 1.00, 95% CI 2-sided [0.63 to 1.37]

3. Secondary Outcome: Change From Baseline in Daily Subject-reported AM and PM rTOSS Averaged Over the Two-week Treatment Period in Participants With a Baseline rTOSS >= 5.0
Description: TOSS is the sum of individual ocular symptoms of itching, tearing, and redness. Subjects assess each individual symptoms on a scale of 0-3 where:
  0 = absent
  1. = mild
  2. = moderate
  3. = severe Therefore, TOSS ranges from 0-9 (with 0 representing an absence of symptoms and higher scores reflecting more severe symptoms). Reflective TOSS symptom scores assess symptoms over the previous 12-hour time interval. Difference was calculated as week two treatment average - baseline. Greater reductions in the change from baseline score indicate greater improvement.
Time Frame: Week 0-2
Population: Intent to treat population. In participants with a baseline rTOSS >= 5.0
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | 80 mcg Ciclesonide | 160 mcg Ciclesonide | Placebo
Number analyzed (Participants) | 164 | 160 | 147
units on a scale | -1.06 (0.12) | -1.05 (0.12) | -0.44 (0.12)
Statistical Analysis 1: Comparison: 80 mcg Ciclesonide vs Placebo; Dmitrienko's tree-structured gatekeeping method was used for multiple comparisons; Test type: Superiority or Other; p = 0.0004, ANCOVA; Mean Difference (Final Values) = 0.61, 95% CI 2-sided [0.28 to 0.95]
Statistical Analysis 2: Comparison: 160 mcg Ciclesonide vs Placebo; Dmitrienko's tree-structured gatekeeping method was used for multiple comparisons; Test type: Superiority or Other; p = 0.0005, ANCOVA; Mean Difference (Final Values) = 0.60, 95% CI 2-sided [0.27 to 0.94]

4. Secondary Outcome: Change From Baseline in Daily Subject-reported AM rTNSS Averaged Over the Two Week Treatment Period
Description: as for outcome 1
Time Frame: Week 0-2
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | 80 mcg Ciclesonide | 160 mcg Ciclesonide | Placebo
Number analyzed (Participants) | 237 | 234 | 234
Units on a scale | -1.45 (0.14) | -1.56 (0.14) | -0.53 (0.14)

5. Secondary Outcome: Change From Baseline in Daily Subject-reported PM rTNSS Averaged Over the Two Week Treatment Period
Description: as for outcome 1
Time Frame: Week 0-2
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | 80 mcg Ciclesonide | 160 mcg Ciclesonide | Placebo
Number analyzed (Participants) | 237 | 234 | 234
Units on a scale | -1.46 (0.14) | -1.60 (0.14) | -0.51 (0.14)

6. Secondary Outcome: Change From Baseline in Daily Subject-reported AM iTNSS Averaged Over the Two Week Treatment Period
Description: TNSS is the sum of individual symptoms of runny nose, sneezing, itchy nose, and nasal congestions. Subjects assess each individual symptoms on a scale of 0-3 where:
  0 = absent
  1. = mild
  2. = moderate
  3. = severe Therefore, rTNSS values range from 0-12 (with 0 representing an absence of symptoms and higher scores reflecting more severe symptoms). Reflective TNSS measures these symptoms over the previous 10 minute time interval. Difference was calculated as the two week treatment average - baseline. Greater reductions in the change from baseline score indicate greater improvement.
Time Frame: Week 0-2
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | 80 mcg Ciclesonide | 160 mcg Ciclesonide | Placebo
Number analyzed (Participants) | 237 | 234 | 234
Units on a scale | -1.32 (0.13) | -1.37 (0.14) | -0.46 (0.14)

7. Secondary Outcome: Change From Baseline in Daily Subject-reported PM iTNSS Averaged Over the Two Week Treatment Period
Description: as for outcome 2
Time Frame: Week 0-2
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | 80 mcg Ciclesonide | 160 mcg Ciclesonide | Placebo
Number analyzed (Participants) | 237 | 234 | 234
Units on a scale | -1.36 (0.14) | -1.55 (0.14) | -0.49 (0.14)

8. Secondary Outcome: Change From Baseline in Daily Subject-reported AM rTOSS Averaged Over the Two Week Treatment Period in Subjects With Baseline rTOSS ≥5.0
Description: as for outcome 3
Time Frame: Week 0-2
Population: In Subjects With Baseline rTOSS ≥5.0
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | 80 mcg Ciclesonide | 160 mcg Ciclesonide | Placebo
Number analyzed (Participants) | 164 | 160 | 147
Units on a scale | -1.03 (0.12) | -0.98 (0.12) | -0.41 (0.13)

9. Secondary Outcome: Change From Baseline in Daily Subject-reported PM rTOSS Averaged Over the Two Week Treatment Period in Subjects With Baseline rTOSS ≥5.0
Description: as for outcome 3
Time Frame: Week 0-2
Population: In Subjects With Baseline rTOSS ≥5.0
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | 80 mcg Ciclesonide | 160 mcg Ciclesonide | Placebo
Number analyzed (Participants) | 164 | 160 | 147
Units on a scale | -1.09 (0.12) | -1.11 (0.12) | -0.47 (0.13)

10. Secondary Outcome: Change From Baseline in Daily Subject-reported AM iTOSS Averaged Over the Two Week Treatment Period in Subjects With Baseline iTOSS ≥5.0
Description: TOSS is the sum of individual ocular symptoms of itching, tearing, and redness. Subjects assess each individual symptoms on a scale of 0-3 where:
  0 = absent
  1. = mild
  2. = moderate
  3. = severe Therefore, TOSS ranges from 0-9 (with 0 representing an absence of symptoms and higher scores reflecting more severe symptoms). Instantaneous TOSS symptom scores assess symptoms over the previous 10 minute time interval. Difference was calculated as week two treatment average - baseline. Greater reductions in the change from baseline score indicate greater improvement.
Time Frame: Week 0-2
Population: In Subjects With Baseline iTOSS ≥5.0
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | 80 mcg Ciclesonide | 160 mcg Ciclesonide | Placebo
Number analyzed (Participants) | 149 | 150 | 133
Units on a scale | -0.96 (0.13) | -0.99 (0.13) | -0.42 (0.13)

11. Secondary Outcome: Change From Baseline in Daily Subject-reported PM iTOSS Averaged Over the Two Week Treatment Period in Subjects With Baseline iTOSS ≥5.0
Description: as for outcome 10
Time Frame: Week 0-2
Population: In Subjects With Baseline iTOSS ≥5.0
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | 80 mcg Ciclesonide | 160 mcg Ciclesonide | Placebo
Number analyzed (Participants) | 149 | 150 | 133
Units on a scale | -1.06 (0.13) | -1.16 (0.13) | -0.36 (0.14)

12. Secondary Outcome: Change From Baseline in Daily Subject Reported AM and PM iTOSS Averaged Over the Two Week Treatment Period in Subjects With Baseline iTOSS ≥5.0
Description: as for outcome 10
Time Frame: Week 0-2
Population: In Subjects With Baseline iTOSS ≥5.0
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | 80 mcg Ciclesonide | 160 mcg Ciclesonide | Placebo
Number analyzed (Participants) | 149 | 150 | 133
Units on a scale | -1.00 (0.12) | -1.07 (0.12) | -0.40 (0.13)

13. Secondary Outcome: Change From Baseline in Daily Subject-reported AM rNSS Averaged Over the Two Week Treatment Period
Description: NSS is the assessment of the individual symptoms of runny nose, sneezing, itchy nose, and nasal congestions. Subjects assess each individual symptoms on a scale of 0-3 where:
  0 = absent
  1. = mild
  2. = moderate
  3. = severe Reflective NSS measures these symptoms over the previous 12-hour time interval. Baseline was the average of the AM and PM responses obtained during the run-in period up to 6 days prior to randomization. Difference was calculated as the two week treatment average - baseline. Greater reductions in the change from baseline score indicate greater improvement.
Time Frame: Week 0-2
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | 80 mcg Ciclesonide | 160 mcg Ciclesonide | Placebo
Number analyzed (Participants) | 237 | 234 | 234
Units on a scale
  Sneezing | -0.39 (0.04) | -0.43 (0.04) | -0.12 (0.04)
  Runny Nose | -0.32 (0.04) | -0.35 (0.04) | -0.13 (0.04)
  Nasal Itching | -0.38 (0.04) | -0.43 (0.04) | -0.17 (0.04)
  Nasal Congestion | -0.35 (0.03) | -0.36 (0.03) | -0.12 (0.03)

14. Secondary Outcome: Change From Baseline in Daily Subject-reported PM rNSS Averaged Over the Two Week Treatment Period
Description: as for outcome 13
Time Frame: Week 0-2
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | 80 mcg Ciclesonide | 160 mcg Ciclesonide | Placebo
Number analyzed (Participants) | 237 | 234 | 234
Units on a scale
  Sneezing | -0.41 (0.04) | -0.46 (0.04) | -0.13 (0.04)
  Runny Nose | -0.32 (0.04) | -0.37 (0.04) | -0.10 (0.04)
  Nasal Itching | -0.38 (0.04) | -0.44 (0.04) | -0.17 (0.04)
  Nasal Congestion | -0.35 (0.04) | -0.35 (0.04) | -0.11 (0.04)

15. Secondary Outcome: Change From Baseline in Daily Subject-reported AM and PM rNSS Averaged Over the Two Week Treatment Period
Description: as for outcome 13
Time Frame: Week 0-2
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | 80 mcg Ciclesonide | 160 mcg Ciclesonide | Placebo
Number analyzed (Participants) | 237 | 234 | 234
Units on a scale
  Sneezing | -0.40 (0.04) | -0.44 (0.04) | -0.12 (0.04)
  Runny Nose | -0.32 (0.04) | -0.36 (0.04) | -0.11 (0.04)
  Nasal Itching | -0.38 (0.04) | -0.43 (0.04) | -0.16 (0.04)
  Nasal Congestion | -0.35 (0.03) | -0.36 (0.03) | -0.11 (0.03)

16. Secondary Outcome: Change From Baseline in Daily Subject-reported AM iNSS Averaged Over the Two Week Treatment Period
Description: NSS is the assessment of the individual symptoms of runny nose, sneezing, itchy nose, and nasal congestions. Subjects assess each individual symptoms on a scale of 0-3 where:
  0 = absent
  1. = mild
  2. = moderate
  3. = severe Instantaneous NSS measures these symptoms over the previous 10 minute time interval. Baseline was the average of the AM and PM responses obtained during the run-in period up to 6 days prior to randomization. Difference was calculated as the two week treatment average - baseline. Greater reductions in the change from baseline score indicate greater improvement.
Time Frame: Week 0-2
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | 80 mcg Ciclesonide | 160 mcg Ciclesonide | Placebo
Number analyzed (Participants) | 237 | 234 | 234
Units on a scale
  Sneezing | -0.33 (0.04) | -0.33 (0.04) | -0.10 (0.04)
  Runny Nose | -0.30 (0.04) | -0.29 (0.04) | -0.09 (0.04)
  Nasal Itching | -0.38 (0.04) | -0.42 (0.04) | -0.16 (0.04)
  Nasal Congestion | -0.31 (0.03) | -0.33 (0.03) | -0.11 (0.03)

17. Secondary Outcome: Change From Baseline in Daily Subject-reported PM iNSS Averaged Over the Two Week Treatment Period
Description: as for outcome 16
Time Frame: Week 0-2
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | 80 mcg Ciclesonide | 160 mcg Ciclesonide | Placebo
Number analyzed (Participants) | 237 | 234 | 234
Units on a scale
  Sneezing | -0.37 (0.04) | -0.43 (0.04) | -0.14 (0.04)
  Runny Nose | -0.30 (0.04) | -0.35 (0.04) | -0.11 (0.04)
  Nasal Itching | -0.35 (0.04) | -0.44 (0.04) | -0.14 (0.04)
  Nasal Congestion | -0.33 (0.04) | -0.33 (0.04) | -0.09 (0.04)

18. Secondary Outcome: Change From Baseline in Daily Subject-reported AM and PM iNSS Averaged Over the Two Week Treatment Period
Description: NSS is the assessment of the individual symptoms of runny nose, sneezing, itchy nose, and nasal congestions. Subjects assess each individual symptoms on a scale of 0-3 where:
  0 = absent
  1. = mild
  2. = moderate
  3. = severe Instantaneous NSS measures these symptoms over the previous 12-hour time interval. Baseline was the average of the AM and PM responses obtained during the run-in period up to 6 days prior to randomization. Difference was calculated as the two week treatment average - baseline. Greater reductions in the change from baseline score indicate greater improvement.
Time Frame: Week 0-2
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | 80 mcg Ciclesonide | 160 mcg Ciclesonide | Placebo
Number analyzed (Participants) | 237 | 234 | 234
Units on a scale
  Sneezing | -0.35 (0.04) | -0.38 (0.04) | -0.12 (0.04)
  Runny Nose | -0.30 (0.04) | -0.33 (0.04) | -0.10 (0.04)
  Nasal Itching | -0.37 (0.04) | -0.43 (0.04) | -0.15 (0.04)
  Nasal Congestion | -0.32 (0.03) | -0.33 (0.03) | -0.33 (0.03)

19. Secondary Outcome: Change From Baseline in Daily Subject-reported AM rOSS Averaged Over the Two Week Treatment Period in Subjects With Baseline rTOSS ≥5.0
Description: OSS is the assessment of the individual symptoms of runny nose, sneezing, itchy nose, and nasal congestions. Subjects assess each individual symptoms on a scale of 0-3 where:
  0 = absent
  1. = mild
  2. = moderate
  3. = severe Therefore, TOSS ranges from 0-9 (with 0 representing an absence of symptoms and 9 reflecting more severe symptoms). Reflective OSS measures these symptoms over the previous 12-hour time interval. Difference was calculated as the two week treatment average - baseline. Greater reductions in the change from baseline score indicate greater improvement.
Time Frame: Week 0-2
Population: In Subjects With Baseline rTOSS ≥5.0
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | 80 mcg Ciclesonide | 160 mcg Ciclesonide | Placebo
Number analyzed (Participants) | 164 | 160 | 147
Units on a scale
  Itching Eyes | -0.36 (0.04) | -0.33 (0.04) | -0.14 (0.04)
  Redness of Eyes | -0.32 (0.04) | -0.31 (0.04) | -0.12 (0.05)
  Tearing Eyes | -0.36 (0.04) | -0.35 (0.04) | -0.16 (0.04)

20. Secondary Outcome: Change From Baseline in Daily Subject-reported PM rOSS Averaged Over the Two Week Treatment Period in Subjects With Baseline rTOSS ≥5.0
Description: as for outcome 19
Time Frame: Week 0-2
Population: In Subjects With Baseline rTOSS ≥5.0
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | 80 mcg Ciclesonide | 160 mcg Ciclesonide | Placebo
Number analyzed (Participants) | 164 | 160 | 147
Units on a scale
  Itching Eyes | -0.34 (0.04) | -0.35 (0.04) | -0.14 (0.04)
  Redness of Eyes | -0.35 (0.05) | -0.34 (0.05) | -0.16 (0.05)
  Tearing Eyes | -0.39 (0.04) | -0.42 (0.04) | -0.16 (0.05)

21. Secondary Outcome: Change From Baseline in Daily Subject-reported and AM and PM rOSS Averaged Over the Two Week Treatment Period in Subjects With Baseline rTOSS ≥5.0
Description: as for outcome 19
Time Frame: Week 0-2
Population: In Subjects With Baseline rTOSS ≥5.0
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | 80 mcg Ciclesonide | 160 mcg Ciclesonide | Placebo
Number analyzed (Participants) | 164 | 160 | 147
Units on a scale
  Itching Eyes | -0.35 (0.04) | -0.34 (0.04) | -0.14 (0.04)
  Redness of Eyes | -0.33 (0.04) | -0.32 (0.04) | -0.14 (0.05)
  Tearing Eyes | -0.38 (0.04) | -0.38 (0.04) | -0.16 (0.04)

22. Secondary Outcome: Change From Baseline in Daily Subject-reported AM iOSS Averaged Over the Two Week Treatment Period in Subjects With Baseline iTOSS ≥5.0
Description: OSS is the assessment of the individual symptoms of runny nose, sneezing, itchy nose, and nasal congestions. Subjects assess each individual symptoms on a scale of 0-3 where:
  0 = absent
  1. = mild
  2. = moderate
  3. = severe Therefore, TOSS ranges from 0-9 (with 0 representing an absence of symptoms and 9 reflecting more severe symptoms). Instantaneous OSS measures these symptoms over the previous 10 minute time interval. Difference was calculated as the two week treatment average - baseline. Greater reductions in the change from baseline score indicate greater improvement.
Time Frame: Week 0-2
Population: In Subjects With Baseline iTOSS ≥5.0
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | 80 mcg Ciclesonide | 160 mcg Ciclesonide | Placebo
Number analyzed (Participants) | 149 | 150 | 133
Units on a scale
  Itching Eyes | -0.33 (0.04) | -0.32 (0.04) | -0.17 (0.05)
  Redness of Eyes | -0.33 (0.05) | -0.32 (0.05) | -0.10 (0.05)
  Tearing Eyes | -0.31 (0.05) | -0.35 (0.05) | -0.13 (0.05)

23. Secondary Outcome: Change From Baseline in Daily Subject-reported PM iOSS Averaged Over the Two Week Treatment Period in Subjects With Baseline iTOSS ≥5.0
Description: as for outcome 22
Time Frame: Week 0-2
Population: In Subjects With Baseline iTOSS ≥5.0
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | 80 mcg Ciclesonide | 160 mcg Ciclesonide | Placebo
Number analyzed (Participants) | 149 | 150 | 133
Units on a scale
  Itching Eyes | -0.34 (0.04) | -0.36 (0.04) | -0.13 (0.05)
  Redness of Eyes | -0.36 (0.05) | -0.38 (0.05) | -0.13 (0.05)
  Tearing Eyes | -0.36 (0.05) | -0.42 (0.05) | -0.10 (0.05)

24. Secondary Outcome: Change From Baseline in Daily Subject-reported AM and PM iOSS Averaged Over the Two Week Treatment Period in Subjects With Baseline iTOSS ≥5.0
Description: as for outcome 22
Time Frame: Week 0-2
Population: In Subjects With Baseline iTOSS ≥5.0
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | 80 mcg Ciclesonide | 160 mcg Ciclesonide | Placebo
Number analyzed (Participants) | 149 | 150 | 133
Units on a scale
  Itching Eyes | -0.34 (0.04) | -0.34 (0.04) | -0.15 (0.04)
  Redness of Eyes | -0.34 (0.04) | -0.35 (0.04) | -0.12 (0.05)
  Tearing Eyes | -0.33 (0.04) | -0.38 (0.04) | -0.12 (0.05)

25. Secondary Outcome: Change From Baseline in Overall Score of the Rhinoconjunctivitis Quality of Life Questionnaire With Standard Activities (RQLQ(S)) in Participants With a Baseline Overall Score >= 3.0
Description: The RQLQ(S) in impaired subjects (baseline RQLQ[S] score ≥3.0) at baseline and end of week 2. It consists of 28 questions, each question measured on a scale of 0-6 where a higher score indicates poor quality of life. Domains: Activities (questions 1-3), Sleep (questions 4-6), Non-Nose/Eye Symptoms (questions 7-13), Practical Problems (questions 14-16), Nasal Symptoms (questions 17-20), Eye Symptoms (questions 21-24), and Emotional (questions 25-28). The overall RQLQ(S) score was calculated as the average of the mean domain scores.
Time Frame: Week 0-2
Population: In participants with a Baseline overall score >= 3.0
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | 80 mcg Ciclesonide | 160 mcg Ciclesonide | Placebo
Number analyzed (Participants) | 186 | 181 | 180
units on a scale | -1.05 (0.10) | -1.07 (0.10) | -0.42 (0.10)

26. Secondary Outcome: Onset of Improvement in Instantaneous Total Nasal Symptoms Scores (iTNSS)
Description: Onset of nasal improvement was defined as the first assessment at which iTNSS for active treatment demonstrated an improvement over placebo from baseline.
  TNSS is the sum of individual symptoms of runny nose, sneezing, itchy nose, and nasal congestions. Subjects assess each individual symptoms on a scale of 0-3 where: 0 = absent, 1 = mild, 2 = moderate, 3 = severe Therefore, iTNSS values range from 0-12 (with 0 representing an absence of symptoms and 12 reflecting more severe symptoms). Instaneous measures these symptoms over the previous 10 minute time interval.
Time Frame: Baseline and up to 36 hours
Population: Intent to Treat Population. Some participants excluded for missing data.
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | 80 mcg Ciclesonide | 160 mcg Ciclesonide | Placebo
Number analyzed (Participants) | 237 | 235 | 235
Units on a scale
  Day 1, 4 Hours Postdose (n=237, 233, 233) | -0.77 (0.15) | -0.79 (0.15) | -0.84 (0.15)
  Day 1, 6 Hours Postdose (n=235, 234, 231) | -1.19 (0.16) | -1.36 (0.16) | -1.19 (0.16)
  Day 1, 8 Hours Postdose (n=236, 233, 233) | -1.31 (0.16) | -1.35 (0.16) | -1.14 (0.16)
  Day 1, 10 Hours Postdose (n=237,232,231) | -1.34 (0.16) | -1.19 (0.16) | -0.90 (0.16)
  Day 1, 12 Hours Postdose (n=236, 233, 233) | -1.14 (0.16) | -1.15 (0.16) | -0.87 (0.16)
  Day 2, Predose (n=237,234,233) | -0.57 (0.15) | -0.81 (0.15) | -0.45 (0.15)
  Day 2, 6 Hours Postdose (n=237,233,231) | -1.56 (0.17) | -1.59 (0.17) | -1.16 (0.17)
  Day 2, 12 Hours Postdose (n=235,233,232) | -1.35 (0.16) | -1.59 (0.17) | -0.77 (0.17)

27. Secondary Outcome: Onset of Improvement in Instantaneous Total Ocular Symptoms Scores (iTOSS) in Subjects With Baseline iTOSS ≥5.0
Description: Onset of improvement iTOSS was defined as the first assessment at which iTOSSS for active treatment demonstrated an improvement over placebo from baseline. TOSS is the sum of individual ocular symptoms of itching, tearing, and redness. Subjects assess each individual symptoms on a scale of 0-3 where:
  0 = absent
  1. = mild
  2. = moderate
  3. = severe Therefore, TOSS ranges from 0-9 (with 0 representing an absence of symptoms and 9 reflecting more severe symptoms). Instantaneous TOSS symptom scores assess symptoms over the previous 10 minute time interval.
Time Frame: Baseline and up to 48 hours
Population: In Subjects With Baseline iTOSS ≥5.0
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | 80 mcg Ciclesonide | 160 mcg Ciclesonide | Placebo
Number analyzed (Participants) | 149 | 150 | 134
Units on a scale
  Day 1, 4 Hours Postdose (n=149, 150, 132) | -0.69 (0.14) | -0.57 (0.14) | -0.53 (0.15)
  Day 1, 6 Hours Postdose (n=149, 150, 132) | -0.93 (0.16) | -0.83 (0.16) | -0.75 (0.17)
  Day 1, 8 Hours Postdose (n=148, 150, 132) | -0.97 (0.15) | -0.97 (0.15) | -0.72 (0.16)
  Day 1, 10 Hours Postdose (n=149, 150, 132) | -1.02 (0.16) | -0.79 (0.15) | -0.69 (0.17)
  Day 1, 12 Hours Postdose (n=149, 148, 132) | -0.80 (0.15) | -0.83 (0.15) | -0.49 (0.16)
  Day 2, Predose (n=149, 149, 132) | -0.29 (0.15) | -0.37 (0.15) | -0.09 (0.16)
  Day 2, 6 Hours Postdose (n=149, 150, 131) | -1.11 (0.16) | -1.15 (0.16) | -0.71 (0.17)
  Day 2, 12 Hours Postdose (n=149, 149, 132) | -1.09 (0.16) | -1.26 (0.16) | -0.47 (0.17)

28. Secondary Outcome: Time to Maximal Effect as Measured by Change From Baseline in the Average AM and PM Reflective Total Nasal Symptoms Scores (rTNSS)
Description: The time to maximal effect is defined as the number of days until the first treatment day on which the estimated difference between Ciclesonide HFA and placebo is at least 90% of the largest estimated difference. This is based on the analyses of change from baseline in the average of AM and PM reflective TNSS scores for each day.
Time Frame: Week 0-2
Population: Intent to Treat Population
Measure: Least Squares Mean (Standard Error); unit: days
Arm/Group | 80 mcg Ciclesonide | 160 mcg Ciclesonide
Number analyzed (Participants) | 237 | 235
days | 13 (0.20) | 8 (0.17)

ADVERSE EVENTS:
Description: A treatment emergent adverse event is defined as an event with onset data occuring on or after the date of first dose of study medication. A subject with multiple events per system organ class or per preferred term was counted only once per system organ class.
Arm/Group | 80 mcg Ciclesonide | 160 mcg Ciclesonide | Placebo
Serious Adverse Events (participants affected / at risk) | 0/237 | 1/235 | 0/235
Other Adverse Events (participants affected / at risk) | 21/237 | 14/235 | 22/235
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 80 mcg Ciclesonide (N=237) | 160 mcg Ciclesonide (N=235) | Placebo (N=235)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 80 mcg Ciclesonide (N=237) | 160 mcg Ciclesonide (N=235) | Placebo (N=235)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 8 (9) | 5 (7) | 10 (11)
Nasal discomort (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 5 (5) | 7 (7)
Nasal septum disorder (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 1 (1) | 3 (3)
Instillation site irritation (General disorders) | 5 (5) | 3 (3) | 2 (2)

LIMITATIONS AND CAVEATS:
This study was not designed or powered for a comparison of the 80mcg dose with the 160mcg dose therefore no statistical comparisons were planned between the two active groups. Publication references to 74 and 148mcg are equivalent to 80 and 160mcg

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other